CLINICAL TRIAL: NCT06213285
Title: Cardiac Computed Tomography Following Watchman FLX Left Atrial APPENDage Closure
Brief Title: APPEND-CT Registry
Acronym: APPEND-CT
Status: Enrolling by invitation | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Mayo Clinic (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Anders Kramer, MD, PhD-fellow, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: ISRCAR00442
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Ischemic; Device Related Thrombosis; Atrial Fibrillation
Keywords: Left Atrial Appendage Occlusion; Cardiac Computed Tomography; Watchman FLX
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Watchman FLX left atrial appendage occlusion — Early (30-120 days) CT follow-up after Watchman FLX LAAO
  Other Names: left atrial appendage closure; LAAO; LAAC

SUMMARY:
The APPEND-CT registry is an investigator-driven multicenter retrospective observational database intended to compile cardiac CT follow-up data after Watchman FLX device implantation and function as a platform for answering clinical and research questions within LAAC follow-up. The derived studies should support therapeutic decision-making, improve risk-stratification in LAAC and help generate hypotheses for potential future clinical intervention trials.

DETAILED DESCRIPTION:
An investigator-driven multicenter retrospective observational database enrolling patients from high-volume North American and European centers. The database will include Watchman FLX implanted patients with a minimum of one follow-up cardiac CT performed within 45-120 days post-procedure. Additional timepoints may be entered. Cardiac CT scans are to be uploaded and will be analyzed by the core-lab at Aarhus University Hospital.

Investigator-reported findings will be systematically reported to the database. This includes information on baseline characteristics, preprocedural planning, implantation details, discharge medication, follow-up imaging and clinical endpoints of interest.

As a minimum, investigator-reported endpoints will be collected from patient registries at one-year follow-up by site-investigators. Endpoints of interest include ischemic stroke, systemic embolism, major bleeding, mortality, device-related thrombosis, pericardial effusion, vascular complications, and device migration.

ELIGIBILITY:
Inclusion Criteria:

* Watchman FLX LAAO
* A minimum of one follow-up cardiac CT performed within 30-120 days post-procedure.
* A minimum of one year clinical follow-up data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Watchman FLX implanted patients with a minimum of one early follow-up cardiac CT.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke | Minimum 12 months
  Clinically affirmed ischemic stroke

SECONDARY OUTCOMES:
Device-related thrombosis | Minimum 12 months
  High-grade hypoattenuated thickening as seen on cardiac CT
Major bleeding | Minimum 12 months
  BARC >=2
All-cause and cardiovascular mortality | Minimum 12 months
  As defined in the Munich consensus

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kramer, MD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Patient data will be registered under a pseudonymous registry-ID and will not be personally identifiable.